CLINICAL TRIAL: NCT06969911
Title: Long-term Performance and Longevity of Minimally Invasive CAD/CAM Versus Conventional Anterior Veneer Restorations: a Randomized Controlled Trial Over 5 Years.
Brief Title: Clinical Evaluation of CAD/CAM vs. Conventional Veneer Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heinrich-Heine University
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-01

CONDITIONS: Malformed Tooth
MeSH Terms: conditions — Tooth Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Conventional veneer restoration (Sham Comparator): Therapeutic intervention with minimally invasive traditionally fabricated all-ceramic anterior veneers.
  Interventions: Procedure: Laminate Veneer Convetional
- Study Group: CAD/CAM veneer restoration (Active Comparator): Therapeutic intervention with minimally invasive CAD/CAM all-ceramic anterior veneers.
  Interventions: Procedure: Laminate veneer CAD/CAM

INTERVENTIONS:
Procedure: Laminate veneer CAD/CAM — Minimally invasive therapeutic intervention with CAD/CAM veneers
  Arms: Study Group: CAD/CAM veneer restoration
Procedure: Laminate Veneer Convetional — Minimally invasive therapeutic intervention with CAD/CAM veneers
  Arms: Control Group: Conventional veneer restoration

SUMMARY:
The aim of the study is to clinically evaluate tooth-supported veneer restorations fabricated using the CAD/CAM process in comparison to conventionally manufactured pressed veneers on anterior teeth and to assess their long-term performance. Survival and success rates of anterior veneer restorations, as well as patient satisfaction, will be evaluated.

DETAILED DESCRIPTION:
Functional and aesthetic complaints caused by congenital malformations and acquired tooth damage are widely spread. Discomfort involves reduced chewing ability, phonetic problems, hypersensitivity and aesthetic impairments.

Conventionally fabricated all-ceramic veneer restorations reveal a long history of clinical success in minimally invasive rehabilitation of the anterior dentition. Nevertheless, conventional manufacturing techniques are prone to fabrication mistakes and must be handled by experienced dental technicians and dentists which results in very high fabrication costs. Therefore, access to minimally invasive restorations is currently restricted for most of the patients. Innovative CAD/CAM techniques have revolutionised restorative treatment options over the last decades and have made all-ceramic restorations more affordable for patients. With further improvements of the CAD/CAM milling devices the machinability of high-strength glass ceramic is now possible.

The aim of both treatment procedures will be to avoid any extensive additional tooth structure removal, to provide long-term survival and success of the integrated restorations and to improve patient´s satisfaction. Up to now scientific evidence on the clinical performance of CAD/CAM fabricated veneers is very limited. Aim of this trial is to evaluate if the clinical performance of anterior restorations after minimally invasive therapeutic intervention with CAD/CAM veneers compared to conventionally fabricated veneers. Functional and aesthetic treatment results will be assessed for five years and evaluated with regard to failure and succes veneer restorations as well as patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients that reveal indication for a minimum of 2 and a maximum of 6 anterior veneer restorations

Exclusion Criteria:

- Patients that reveal multiple missing teeth, poor oral hygiene, pronounced parafunctions or with allergies to any of the applied materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Prosthetic survival time | 5 Years
  The primary objective is to compare the prosthetic survival time of the restorations (conventional vs. CAD/CAM veneers).

SECONDARY OUTCOMES:
Prosthetic success | 5 Years
  The secondary objectives are to compare the prosthetic success of the restorations (conventional vs. CAD/CAM veneers), the documentation of failures such as fractures and the assessment of patient centered satisfaction.

IPD SHARING:
Plan to Share IPD: No